CLINICAL TRIAL: NCT01686347
Title: Epidural Analgesia and Troubles of Fetal Cardiaq Rythm : Effect of the Systemic Transfer of Ropivacaine and Sufentanil
Acronym: epidarc
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2010/146/HP
Record Dates: First submitted 2012-06-07; First posted 2012-09-18 (Estimated); Last update posted 2016-01-25 (Estimated); Status verified 2016-01

CONDITIONS: Fetal Cardiac Rhythm Abnormalities
Keywords: epidural analgesia; fetal cardiac rythm; ropivacaine; sufentanil
MeSH Terms: interventions — Ropivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- fetal cardiac rhythm abnormally (Other): patient at term, in spontanous labor with fetal cardiac rythm abnormally which occurs 30 minutes after the epidural analgesia induction
  Interventions: Drug: ropivacaine
- control group (Other): patient at term, spontaneous labor, without any fetal cardiac rhythm abnormalies during the 30 minutes after the epidural analgesia induction
  Interventions: Drug: ropivacaine

INTERVENTIONS:
Drug: ropivacaine

SUMMARY:
The aim of the investigators study is to demonstrate the association between fetal cardiac rhythm abnormalies after epidural analgesia and the maternal systemic transfer of ropivacaine and/or sufentanil.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or more
* nulliparous

  _ one fetus
* head first
* spontaneous labor
* epidural analgesia
* no fetal cardiac rhythm abnormalies before the epidural analgesia
* no active management of labor during 30 minutes after the epidural analgesia induction
* at term
* signature of the consent form

Exclusion Criteria:

* pathological pregnancy
* low maternal blood pressure during the 30 minutes after the epidural analgesia
* uterin contraction which last for 5 minutes or more
* more than 6 uterin contractions during a 10 minutes period
* Ropivacaine contraindication
* sufentanil contraindication

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-06; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Plasmatic concentrations compared maternal ropivacaine based on the presence of abnormal fetal heart rate | 1 day
  Maternal Plasmatic concentrations of ropivacaine will be measured in mg / liter of maternal blood and the median of each group will be compared by paired Wilcoxon test

SECONDARY OUTCOMES:
Plasmatic concentrations compared maternal sufentanil based on the presence of abnormal fetal heart rate | 1 day
  Maternal Plasmatic concentrations of sufentanil will be measured in mg / liter of maternal blood and the median of each group will be compared by paired Wilcoxon test

CONTACTS AND LOCATIONS:
Locations (1):
- centre hospitalier universitaire de Rouen, Hopital Charles Nicolle, Rouen, France